CLINICAL TRIAL: NCT02457325
Title: Comparative Analysis Between 2% and Articaine Articaine 4%, Both With 1: 200,000 Epinephrine: Evaluation of Anesthetics Efficacy, Intraoperative Bleeding and Hemodynamic Parameters in Extraction of Lower Third Molars
Brief Title: Lower Third Molar Removal With 2% and 4% Articaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carlos Ferreira dos Santos, PhD, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: U1111-1120-3074
Record Dates: First submitted 2015-05-18; First posted 2015-05-29 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Impacted Third Molar Tooth; Adverse Reaction to Other Local Anesthetics
Keywords: Articaine; Lower third molar; Oral Surgery
MeSH Terms: interventions — Surgical Procedures, Operative; Carticaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery With 2% Articaine first, then Surgery With 4%Articaine (Experimental): First Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne)
  Interventions: Drug: Surgery with 2%Articaine first, then Surgery with 4% Articaine
- Surgery With 4%Articaine first, then Surgery With 2% Articaine (Experimental): First Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne)
  Interventions: Drug: Surgery with 4%Articaine first, then Surgery with 2% Articaine

INTERVENTIONS:
Drug: Surgery with 2%Articaine first, then Surgery with 4% Articaine — First Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne)
  Other Names: Lower third molar with 2% Articaine and 4% Articaine
  Arms: Surgery With 2% Articaine first, then Surgery With 4%Articaine
Drug: Surgery with 4%Articaine first, then Surgery with 2% Articaine — First Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne)
  Other Names: Lower third molar with 4% Articaine and 2% Articaine
  Arms: Surgery With 4%Articaine first, then Surgery With 2% Articaine

SUMMARY:
The present clinical trial randomized compared the clinical efficacy of the local anesthetics articaine in two concentrations, 2% and 4%, in association with 1:200,000 adrenaline, for the removal of lower third molars. Onset, duration of postoperative analgesia, duration of anesthetic action on soft tissues, intraoperative bleeding, hemodynamic parameters, postoperative mouth opening and wound healing at the 7th postoperative day were evaluated. For this purpose, 50 healthy volunteers underwent removal of symmetrically positioned lower third molars, in two separate appointments (one to two months apart), under local anesthesia with either articaine 2% or 4% (both with 1:200,000 adrenaline) in a double-blind, randomized and crossed manner.

DETAILED DESCRIPTION:
The present clinical trial randomized compared the clinical efficacy of the local anesthetics articaine in two concentrations, 2% and 4%, in association with 1:200,000 adrenaline, for the removal of lower third molars. Onset, duration of postoperative analgesia, duration of anesthetic action on soft tissues, intraoperative bleeding, hemodynamic parameters, postoperative mouth opening and wound healing at the 7th postoperative day were evaluated. This study evaluated the clinical efficacy of two concentrations (2% and 4%) of the local anesthetic articaine, a local anesthetic of moderate duration, associated with adrenalin at 1: 200,000 in 50 patients aged less than 18 years and in need of extraction of the two third molars with similar positions. Evaluated the following parameters: 1) onset of action of the anesthetic agent, 2) the total amount of anesthesia used during surgery, 3) onset and duration of surgery after the administration of the local anesthetic, 4) the incidence, type and severity of adverse reactions, 5) postoperative control of mouth opening, 6) subjective evaluation of postoperative pain, 7) postoperative duration of anesthesia, 8) Total amount of relief medication and 9) heart rate and systolic and diastolic blood pressure before during and after surgery. The comparative analysis of the data and the application of proper statistical tests provided the basis for an assessment of the efficiency of both concentrations of the local anesthetic articaine (2% and 4%) with adrenalin at 1: 200,000.

ELIGIBILITY:
Inclusion Criteria:

* Need of lower third molar surgeries in similar positions

Exclusion Criteria:

* Presence of systemic diseases;
* Presence of local inflammation and/or infection;
* Any history of allergic reaction to local anesthetics, gastrointestinal bleeding or ulceration;
* Cardiovascular and kidney diseases;
* Asthma and allergy to aspirin, piroxicam or any other non-steroidal antiinflammatory drug;
* Regular use of any non-steroidal antiinflammatory drug, pregnancy or breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos F Santos, PhD, Principal Investigator — Bauru School of Dentistry/University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No
Data are presented as mean and standard deviation

REFERENCES:
- [Derived] Senes AM, Calvo AM, Colombini-Ishikiriama BL, Goncalves PZ, Dionisio TJ, Sant'ana E, Brozoski DT, Lauris JR, Faria FA, Santos CF. Efficacy and Safety of 2% and 4% Articaine for Lower Third Molar Surgery. J Dent Res. 2015 Sep;94(9 Suppl):166S-73S. doi: 10.1177/0022034515596313. Epub 2015 Jul 22. PMID 26202994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients were recruited to perform bilateral surgery for extraction of lower third molars, at the Faculty of Dentistry of Bauru
Pre-assignment Details: 46 of 50 patients were randomized. Of those not randomized, 4 did not return to folow up and were excluded of the study.
Groups:
- Surgery With 2% Articaine First, Then 4% Articaine: First Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne)
- Surgery With 4%Articaine First, Then 2% Articaine: First Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne)
Period: First Intervention (1 Day)
Arm/Group | Surgery With 2% Articaine First, Then 4% Articaine | Surgery With 4%Articaine First, Then 2% Articaine
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: Washout (1-2 Months)
Arm/Group | Surgery With 2% Articaine First, Then 4% Articaine | Surgery With 4%Articaine First, Then 2% Articaine
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Surgery With 2% Articaine First, Then 4% Articaine | Surgery With 4%Articaine First, Then 2% Articaine
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgery With 4%Articaine First, Then Surgery With 2%Articaine: First Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne), Washout (1-2 months), and Second Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne)
- Total: Total of all reporting groups
Arm/Group | Surgery With 2%Articaine First, Then Surgery With 4% Articaine | Surgery With 4%Articaine First, Then Surgery With 2%Articaine | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 23 [18 to 44] | 23 [18 to 44] | 23 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  Brazil | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Onset of Anesthetic
Description: Onset of anesthetic agent action, as determined by the loss of sensibility of the inferior lip, the corresponding half of the tongue, and the mucosa as reported by the patient.
Time Frame: During the surgical procedure, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Surgery With 2%Articaine: Intervention (1 day - third molar surgery with infiltration of one cartridge of 2% articaíne)
- Surgery With 4%Articaine: Intervention (1 day - third molar surgery with infiltration of one cartridge of 4% articaíne)
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
minutes | 1.5 (0.6) | 1.5 (0.6)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.192, t-test, 2 sided

2. Primary Outcome: Quality of Anesthesia
Description: Quality of anesthesia during surgery based on a category 3-point scale: 1) the patient reported no discomfort; 2) the patient reported discomfort, without the need to supplement the anesthesia; 3) reported some discomfort by the patient, requiring anesthesia complementation. Intraoral bleeding that will be evaluated by the surgeon according to a 3-point scale (1: minimal, 2: normal and 3: Maximum), immediately after the following steps: injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing.
Time Frame: During the surgical procedure, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
units on a scale | 1.8 (1.0) | 1.8 (1.0)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.457, t-test, 2 sided

3. Primary Outcome: Intraoperative Bleeding
Description: Intraoperative bleeding, rated by the surgeon according to a 3-point category rating scale (1-minimal bleeding; 2-normal bleeding; 3-excessive bleeding) (SISK, 1986), immediately after the following steps: injection of the first cartridge of articaine, tissue incision, flap reflection, bone removal (when this procedure was necessary), tooth extraction, cleaning of the operated site, and completion of suturing.
Time Frame: During the surgical procedure, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
units on a scale | 1.1 (0.1) | 1.1 (0.2)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine; Test type: Superiority or Other; p = 0.158, t-test, 2 sided

4. Primary Outcome: Blood Pressure
Description: mean blood pressure was verified and recorded at surgical moments previously described (injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing), carried out with the aid of a system for monitoring hemodynamic parameters.
Time Frame: During the surgical procedure, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
mmHg | 119 (11) | 123 (11)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.953, t-test, 2 sided

5. Primary Outcome: Heart Rate
Description: Heart rate to be verified and recorded surgical at moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.
Time Frame: During the surgical procedure, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
bpm | 73 (17) | 73 (17)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.693, t-test, 2 sided

6. Primary Outcome: Oxygen Saturation
Description: Oxygen saturation to be verified and recorded at surgical moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.
Time Frame: During the surgical procedure, an average of 30 minutes
Measure: Mean (Standard Deviation); unit: percentage of oxigen in blood
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
percentage of oxigen in blood | 99 (4) | 99 (1)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.158, t-test, 2 sided

7. Secondary Outcome: Duration of Post-operative Analgesia
Description: Duration of post-operative analgesia (in minutes) provided by the local anesthetic will be determined by the difference between the end time of the completion of suture and the one for the first intake piroxicam capsule for the relief of discomfort after surgery, the patient noted in token that you will be provided. Duration of post-surgical anesthesia (in minutes) on the soft tissues provided by local anesthetic, represented by the lack of sensitivity in the mucosa, tongue and lower lip after the surgery. The patient will note the time at which this phenomenon happens on the card which will be provided.
Time Frame: During the day of the surgery, 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
minutes | 133 (110) | 125 (102)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.192, t-test, 2 sided

8. Secondary Outcome: Postoperative Mouth Opening
Description: Mouth opening (mm) between the mesial-incisal corners of the upper and lower right central incisors at maximum opening of the jaws was measured and recorded. Results presented below represent those assessed on the seventh postoperative day.
Time Frame: Seventh postoperative days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
mm | 36 (10) | 35 (11)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.512, t-test, 2 sided

9. Secondary Outcome: Wound Healing of the Operated Area
Description: Quality of wound healing of the operated area classified by the surgeon according to a scale of three types of points: 1-normal healing, 2-delayed healing, 3-wound healing complicated by the presence of alveolitis at the time of removal of the suture (7th postoperative day).
Time Frame: Seventh postoperative day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
units on a scale | 1.2 (0.4) | 1.4 (0.6)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.115, t-test, 2 sided

10. Secondary Outcome: Evaluation of Post-surgical Pain
Description: Subjective evaluation of post-surgical pain, which was annotated by the volunteer, a Visual Analogue Scale (VAS, 0-100 mm - higher values represent a worse outcome) in the postoperative period.
Time Frame: Seventh postoperative day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
units on a scale | 26 (29) | 26 (29)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.730, t-test, 2 sided

11. Secondary Outcome: Postoperative Anesthesia
Description: Duration of postoperative anesthesia, represented by the lack of sensibility of the mucosa, tongue, and inferior lip.
Time Frame: During the day of the surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Number analyzed (Participants) | 46 | 46
minutes | 187 (90) | 215 (77)
Statistical Analysis 1: Comparison: Surgery With 2%Articaine vs Surgery With 4%Articaine; Test type: Superiority or Other; p = 0.835, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month after surgery
Arm/Group | Surgery With 2%Articaine | Surgery With 4%Articaine
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 1/46 | 1/46
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery With 2%Articaine (N=46) | Surgery With 4%Articaine (N=46)
paresthesia of the lingual nerve (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Temporary paresthesia of lingual nerve (3 months) on both sides of surgeries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes